CLINICAL TRIAL: NCT02632175
Title: A Multi-Center, Open-Label Study of the Human Anti-TNF Monoclonal Antibody Adalimumab to Evaluate Long-Term Safety and Tolerability of Repeated Administration of Adalimumab in Pediatric Subjects With Ulcerative Colitis Who Completed the Study M11-290
Brief Title: Long-term Safety and Efficacy Study of Adalimumab in Pediatric Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-870; 2015-001346-29 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects receiving Adalimumab (Experimental): Subjects receiving Adalimumab up to 288 weeks
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — every other week or weekly subcutaneous injection

SUMMARY:
This study assesses the long-term safety and efficacy of adalimumab in pediatric subjects with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

- Subject must have successfully enrolled and completed M11-290 study

Exclusion Criteria:

- Subject considered by the investigator, for any reason, to be an unsuitable candidate

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (16):
- United States (4):
  - Arnold Palmer Hospital /ID# 147295, Orlando, Florida
  - MNGI Digestive Health, P. A. /ID# 147294, Minneapolis, Minnesota
  - Mayo Clinic - Rochester /ID# 147304, Rochester, Minnesota
  - MultiCare Institute Health System /ID# 169005, Tacoma, Washington
- Japan (3):
  - Kurume University Hospital /ID# 145710, Kurume-shi, Fukuoka
  - Juntendo University Hospital /ID# 147315, Bunkyo-ku, Tokyo
  - National Center for Child Health and Development /ID# 147312, Setagaya-ku, Tokyo
- Poland (5):
  - Uniwersytecki Szpital Dzieciecy w Krakowie /ID# 147279, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego /ID# 147310, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM /ID# 147280, Warsaw, Masovian Voivodeship
  - Gabinet Lekarski Bartosz Korcz /ID# 147281, Rzeszów, Podkarpackie Voivodeship
  - Instytut Centrum Zdrowia Matki Polki /ID# 169017, Lodz, Łódź Voivodeship
- Univerzitna nemocnica Martin /ID# 147283, Martin, Žilina Region, Slovakia
- Hospital Universitario Vall d'Hebron /ID# 147288, Barcelona, Spain
- United Kingdom (2):
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 147290, London, Greater London
  - Duplicate_The Royal Free London NHS Foundation Trust /ID# 147292, London, Greater London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This Clinical Study maybe evaluating a usage that is not currently FDA-approved. Please see US prescribing information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants received adalimumab every other week (EOW) or every week (EW) subcutaneous injection for up to 288 weeks.
  (Prior to Amendment 4): Participants who enrolled into the study from blinded treatment in Study M11-290 received open-label adalimumab 0.6 mg/kg (maximum dose of 40 mg) EOW.
  Participants who received open-label adalimumab 0.6 mg/kg (maximum of 40 mg) EW in Study M11-290 maintained the same dose in Study M10-870.
  (After Amendment 4): Participants with a body weight < 25 kg received open-label adalimumab 20 mg EOW.
  Participants with a body weight ≥ 25 kg - < 40 kg received open-label adalimumab 40 mg EOW.
  Participants with a body weight ≥ 40 kg received open-label adalimumab 80 mg EOW.
Period: Overall Study
Arm/Group | Adalimumab
Started | 59
Completed | 28
Not Completed | 31
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 18
Not completed — Required alternative (or prohibited) therapy | 1
Not completed — Subject noncompliance | 3
Not completed — other | 2

BASELINE CHARACTERISTICS:
Population: Integrated Full Analysis Set (IFAS) included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (3.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Proportion of Participants with Partial Mayo Score (PMS) Remission at Baseline [Count of Participants; unit: Participants] — The Partial Mayo Score (PMS) is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Physician's Global Assessment (PGA), scored from 0 (normal) to 3 (severe disease).
  The overall Partial Mayo score ranges from 0 to 9 with higher scores representing more severe disease.
  Participants | 46
Proportion of Participants with PMS Response at Study M11-290 Baseline [Count of Participants; unit: Participants] — The Partial Mayo Score (PMS) is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Physician's Global Assessment (PGA), scored from 0 (normal) to 3 (severe disease).
  The overall Partial Mayo score ranges from 0 to 9 with higher scores representing more severe disease.
  Participants | 54
Proportion of Participants Who Achieve PUCAI Remission at Baseline [Count of Participants; unit: Participants] — The Pediatric Ulcerative Colitis Activity Index (PUCAI) measures UC disease activity in children and adolescents by evaluating the following 6 areas: abdominal pain, number of stools per day, stool consistency, amount of blood in stools, nocturnal stooling, and activity level.
  The PUCAI score ranges from 0 to 85 with higher scores representing more severe disease.
  Recommended cut-off scores to differentiate disease activity are 0-9 (inactive), 10-34 (mild), 35-64 (moderate), and > 65 (severe).
  Participants | 42
Proportion of Participants Who Achieve PUCAI Response at Study M11-290 Baseline [Count of Participants; unit: Participants] — The Pediatric Ulcerative Colitis Activity Index (PUCAI) measures UC disease activity in children and adolescents by evaluating the following 6 areas: abdominal pain, number of stools per day, stool consistency, amount of blood in stools, nocturnal stooling, and activity level.
  The PUCAI score ranges from 0 to 85 with higher scores representing more severe disease.
  Recommended cut-off scores to differentiate disease activity are 0-9 (inactive), 10-34 (mild), 35-64 (moderate), and > 65 (severe).
  Participants | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 70 days following last dose of study drug (up to 298 weeks).
Population: Integrated Full Analysis Set (IFAS) included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
Participants
  Any TEAE | 55
  TESAE | 15

2. Primary Outcome: Proportion of Participants Who Achieve Clinical Remission as Measured by Partial Mayo Score (PMS)
Description: The Partial Mayo Score (PMS) is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Physician's Global Assessment (PGA), scored from 0 (normal) to 3 (severe disease).
  The overall Partial Mayo score ranges from 0 to 9 with higher scores representing more severe disease.
  Clinical remission was defined as a PMS ≤ 2 and no individual subscore > 1.
Time Frame: Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96,108,120, 144, 168, 192, 216, 240, 264, and 288
Population: Integrated Full Analysis Set (IFAS) included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
Participants
  Week 4: number analyzed (Participants) | 58
  Week 4 | 50
  Week 8 | 47
  Week 12 | 51
  Week 24: number analyzed (Participants) | 58
  Week 24 | 43
  Week 36: number analyzed (Participants) | 56
  Week 36 | 45
  Week 48: number analyzed (Participants) | 53
  Week 48 | 40
  Week 60: number analyzed (Participants) | 50
  Week 60 | 42
  Week 72: number analyzed (Participants) | 49
  Week 72 | 42
  Week 84: number analyzed (Participants) | 47
  Week 84 | 40
  Week 96: number analyzed (Participants) | 45
  Week 96 | 36
  Week 108: number analyzed (Participants) | 42
  Week 108 | 37
  Week 120: number analyzed (Participants) | 41
  Week 120 | 33
  Week 144: number analyzed (Participants) | 39
  Week 144 | 32
  Week 168: number analyzed (Participants) | 35
  Week 168 | 31
  Week 192: number analyzed (Participants) | 32
  Week 192 | 30
  Week 216: number analyzed (Participants) | 32
  Week 216 | 29
  Week 240: number analyzed (Participants) | 30
  Week 240 | 28
  Week 264: number analyzed (Participants) | 28
  Week 264 | 27
  Week 288: number analyzed (Participants) | 27
  Week 288 | 25

3. Primary Outcome: Proportion of Participants Who Achieve Clinical Response as Measured by PMS (From Study M11-290 Baseline)
Description: The Partial Mayo Score (PMS) is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Physician's Global Assessment (PGA), scored from 0 (normal) to 3 (severe disease).
  The overall Partial Mayo score ranges from 0 to 9 with higher scores representing more severe disease.
  Clinical response was defined as a decrease in PMS ≥ 2 points and ≥ 30% from Study M11-290 Baseline.
Time Frame: Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96,108,120, 144, 168, 192, 216, 240, 264, and 288
Population: Integrated Full Analysis Set (IFAS) included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
Participants
  Week 4: number analyzed (Participants) | 58
  Week 4 | 56
  Week 8 | 55
  Week 12 | 56
  Week 24: number analyzed (Participants) | 58
  Week 24 | 51
  Week 36: number analyzed (Participants) | 56
  Week 36 | 50
  Week 48: number analyzed (Participants) | 53
  Week 48 | 47
  Week 60: number analyzed (Participants) | 50
  Week 60 | 46
  Week 72: number analyzed (Participants) | 49
  Week 72 | 44
  Week 84: number analyzed (Participants) | 47
  Week 84 | 43
  Week 96: number analyzed (Participants) | 45
  Week 96 | 42
  Week 108: number analyzed (Participants) | 42
  Week 108 | 40
  Week 120: number analyzed (Participants) | 41
  Week 120 | 39
  Week 144: number analyzed (Participants) | 39
  Week 144 | 35
  Week 168: number analyzed (Participants) | 35
  Week 168 | 35
  Week 192: number analyzed (Participants) | 32
  Week 192 | 32
  Week 216: number analyzed (Participants) | 32
  Week 216 | 30
  Week 240: number analyzed (Participants) | 30
  Week 240 | 29
  Week 264: number analyzed (Participants) | 28
  Week 264 | 28
  Week 288: number analyzed (Participants) | 27
  Week 288 | 26

4. Primary Outcome: Proportion of Participants Who Achieve Pediatric Ulcerative Colitis Activity Index (PUCAI) Remission
Description: The Pediatric Ulcerative Colitis Activity Index (PUCAI) measures UC disease activity in children and adolescents by evaluating the following 6 areas: abdominal pain, number of stools per day, stool consistency, amount of blood in stools, nocturnal stooling, and activity level.
  The PUCAI score ranges from 0 to 85 with higher scores representing more severe disease.
  Recommended cut-off scores to differentiate disease activity are 0-9 (inactive), 10-34 (mild), 35-64 (moderate), and > 65 (severe).
  Clinical remission was defined as a PUCAI score < 10.
Time Frame: Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96,108,120, 144, 168, 192, 216, 240, 264, and 288
Population: Integrated Full Analysis Set (IFAS) included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
Participants
  Week 4: number analyzed (Participants) | 58
  Week 4 | 50
  Week 8 | 46
  Week 12 | 50
  Week 24: number analyzed (Participants) | 58
  Week 24 | 42
  Week 36: number analyzed (Participants) | 56
  Week 36 | 44
  Week 48: number analyzed (Participants) | 53
  Week 48 | 39
  Week 60: number analyzed (Participants) | 50
  Week 60 | 38
  Week 72: number analyzed (Participants) | 49
  Week 72 | 42
  Week 84: number analyzed (Participants) | 47
  Week 84 | 40
  Week 96: number analyzed (Participants) | 45
  Week 96 | 37
  Week 108: number analyzed (Participants) | 42
  Week 108 | 37
  Week 120: number analyzed (Participants) | 41
  Week 120 | 34
  Week 144: number analyzed (Participants) | 39
  Week 144 | 33
  Week 168: number analyzed (Participants) | 35
  Week 168 | 30
  Week 192: number analyzed (Participants) | 32
  Week 192 | 28
  Week 216: number analyzed (Participants) | 32
  Week 216 | 28
  Week 240: number analyzed (Participants) | 30
  Week 240 | 27
  Week 264: number analyzed (Participants) | 28
  Week 264 | 26
  Week 288: number analyzed (Participants) | 27
  Week 288 | 24

5. Primary Outcome: Proportion of Participants Who Achieve PUCAI Response (From Study M11-290 Baseline)
Description: The Pediatric Ulcerative Colitis Activity Index (PUCAI) measures UC disease activity in children and adolescents by evaluating the following 6 areas: abdominal pain, number of stools per day, stool consistency, amount of blood in stools, nocturnal stooling, and activity level.
  The PUCAI score ranges from 0 to 85 with higher scores representing more severe disease.
  Recommended cut-off scores to differentiate disease activity are 0-9 (inactive), 10-34 (mild), 35-64 (moderate), and > 65 (severe).
  PUCAI response was defined as a decrease in PUCAI score ≥ 20 points from Study M11-290 Baseline.
Time Frame: Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96,108,120, 144, 168, 192, 216, 240, 264, and 288
Population: Integrated Full Analysis Set (IFAS) included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
Participants
  Week 4: number analyzed (Participants) | 58
  Week 4 | 47
  Week 8 | 47
  Week 12 | 49
  Week 24: number analyzed (Participants) | 58
  Week 24 | 42
  Week 36: number analyzed (Participants) | 56
  Week 36 | 43
  Week 48: number analyzed (Participants) | 53
  Week 48 | 38
  Week 60: number analyzed (Participants) | 50
  Week 60 | 39
  Week 72: number analyzed (Participants) | 49
  Week 72 | 40
  Week 84: number analyzed (Participants) | 47
  Week 84 | 37
  Week 96: number analyzed (Participants) | 45
  Week 96 | 37
  Week 108: number analyzed (Participants) | 42
  Week 108 | 36
  Week 120: number analyzed (Participants) | 41
  Week 120 | 34
  Week 144: number analyzed (Participants) | 39
  Week 144 | 32
  Week 168: number analyzed (Participants) | 35
  Week 168 | 30
  Week 192: number analyzed (Participants) | 32
  Week 192 | 27
  Week 216: number analyzed (Participants) | 32
  Week 216 | 25
  Week 240: number analyzed (Participants) | 30
  Week 240 | 26
  Week 264: number analyzed (Participants) | 28
  Week 264 | 23
  Week 288: number analyzed (Participants) | 27
  Week 288 | 21

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment up to 298 weeks, median time on follow up (median time subjects were followed) was 1723.0 days for adalimumab. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 70 days after the last dose of study drug; mean duration on study drug was 1354.2 days for adalimumab.
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 16/59
Other Adverse Events (participants affected / at risk) | 54/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 5 (6)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 2 (2)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
LATENT TUBERCULOSIS (Infections and infestations) | 1 (1)
LYMPH NODE ABSCESS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
GROWTH FAILURE (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
HAEMATOCOLPOS (Reproductive system and breast disorders) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 7 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (4)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 20 (26)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 3 (4)
GASTRITIS (Gastrointestinal disorders) | 3 (3)
HAEMATOCHEZIA (Gastrointestinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 5 (6)
VOMITING (Gastrointestinal disorders) | 3 (3)
FATIGUE (General disorders) | 3 (4)
PYREXIA (General disorders) | 5 (6)
SEASONAL ALLERGY (Immune system disorders) | 5 (5)
BRONCHITIS (Infections and infestations) | 5 (6)
COVID-19 (Infections and infestations) | 10 (13)
HERPES ZOSTER (Infections and infestations) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 13 (21)
PHARYNGITIS (Infections and infestations) | 8 (9)
TONSILLITIS (Infections and infestations) | 3 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 (26)
URINARY TRACT INFECTION (Infections and infestations) | 4 (7)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9)
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 10 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (9)
HEADACHE (Nervous system disorders) | 9 (11)
DEPRESSION (Psychiatric disorders) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 4 (5)
ACNE (Skin and subcutaneous tissue disorders) | 5 (6)
DERMATITIS (Skin and subcutaneous tissue disorders) | 3 (5)
RASH (Skin and subcutaneous tissue disorders) | 4 (5)
URTICARIA (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT02632175/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02632175/SAP_001.pdf